CLINICAL TRIAL: NCT06738602
Title: Comparison Between Progestin Primed Ovarian Stimulation Protocol and Antagonist Protocol in Hyper-responder Patients Schaduled for Freeze All Policy
Brief Title: Difference Between Progestin Primed Ovarian Stimulation Protocol and Antagonist Protocol
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mostafa Ahmed, Comparison between progestin primed ovarian stimulation protocol and antagonist protocol in hyper-responder patients schaduled for freeze all policy, Assiut University
Other Study IDs: Induction protocols in IVF
Record Dates: First submitted 2024-12-10; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Infertility Assisted Reproductive Technology
Keywords: progestin primed ovarian stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Progestin Primed Ovarian Stimulation Protocol group
- Antagonist Protocol group

SUMMARY:
compare the effectiveness and safety of the progestin primed ovarian stimulation (PPOS) protocol versus the antagonist protocol in hyper-responder patients scheduled for a freeze-all policy

DETAILED DESCRIPTION:
Infertility treatments have evolved significantly over the past few decades, with various protocols being developed to optimize ovarian stimulation in assisted reproductive technology (ART). Among these protocols, the progestin-primed ovarian stimulation (PPOS) and the antagonist protocols have gained prominence, especially in hyper-responders who are scheduled for a freeze-all policy. Hyper-responders are patients who produce an excessive number of eggs in response to ovarian stimulation, which increases the risk of ovarian hyperstimulation syndrome (OHSS), a potentially severe complication .

The PPOS protocol involves the administration of progestins to suppress the premature luteinizing hormone (LH) surge during ovarian stimulation, thereby providing a controlled environment for follicle development. This method has been found to be effective in reducing the risk of OHSS and improving clinical outcomes . On the other hand, the antagonist protocol employs gonadotropin-releasing hormone (GnRH) antagonists to prevent the LH surge, offering a more immediate suppression compared to progestins .

A freeze-all policy, where all viable embryos are frozen for future use rather than being transferred immediately, is often recommended for hyper-responders to further minimize the risk of OHSS . This approach allows for the transfer of embryos in a more physiologically normal uterine environment, potentially improving implantation rates and pregnancy outcomes .

This study aims to compare the effectiveness and safety of the PPOS protocol versus the antagonist protocol in hyper-responder patients scheduled for a freeze-all policy. By examining outcomes such as the number of retrieved oocytes, incidence of OHSS, and pregnancy rates, this research seeks to provide insights into the optimal ovarian stimulation strategy for this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

• All hyper responder patients according to Olivera equation for overian response peridiction index

Exclusion Criteria:

* All normal and poor responder patients according to Olivera equation for overian response peridiction index.
* Sever male factor infertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female with primary or secondary infertility
Study Population: * Eligible patients will be identified and recruited from the IVF Unit at Women's Health Hospital.
  * Informed consent will be obtained from all participants prior to inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
• Clinical pregnancy rate: The presence of a gestational sac with fetal heartbeat on ultrasound at 7 weeks of gestation. • Live birth rate: The delivery of a live-born infant beyond 24 weeks of gestation | 1 year
  the measure unit is the presence of pulsation in 7-week gestational sac or delivery if fetus beyond 24 weeks as if fetus below 24 w gestation , it's considered abortion